CLINICAL TRIAL: NCT05547100
Title: A Phase 1, Open-Label Study of the Breast Milk Pharmacokinetics of Olanzapine and Samidorphan in Healthy Lactating Women
Brief Title: Study of the Breast Milk Pharmacokinetics of Olanzapine and Samidorphan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALKS 3831-112
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Focus of Study is on Healthy Lactating Women
Keywords: Samidorphan; Healthy Lactating Women; LYBALVI; ALKS 3831; Breast milk
MeSH Terms: interventions — lybalvi; Olanzapine; 3-carboxamido-4-hydroxynaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5mg OLZAPINE /10mg SAMIDORPHAN (Experimental): Open label, single dose 5mg OLZ/10 mg SAM
  Interventions: Drug: LYBALVI

INTERVENTIONS:
Drug: LYBALVI — 5 mg Olanzapine/10 mg Samidorphan dose approved for use in treatment for schizophrenia and bipolar I disorder
  Other Names: Olanzapine/samidorphan (OLZ/SAM); ALKS 3831

SUMMARY:
This clinical lactation study is to provide information regarding the PK and amount of OLZ/SAM in breast milk and estimated infant exposure.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥18 and <35 kg/m2
* Subject is lactating, at least 4 weeks post-partum at dosing, and is using or willing to use an electronic breast pump for sample collection
* Subject is willing to temporarily discontinue breastfeeding for the duration of at least 11 days post-dose
* Subject is exclusively breastfeeding and/or pumping milk, or if not exclusively breastfeeding/pumping, has an adequate milk supply as judged by the Investigator
* Subject's infant is able to bottle-feed
* Subject agrees to use contraception during the study

Exclusion Criteria:

* Subject has a history of lumpectomy, mastectomy, breast implants, breast augmentation, or breast reduction surgery
* Breastfeeding is not well-established or milk supply is low as judged by the Investigator
* Subject has mastitis or other condition that may prevent the collection of milk from one or both breasts
* Subject is pregnant or plans to become pregnant during the study
* Subject has had a clinically significant illness within 30 days or has had a serious infection (eg, pneumonia or septicemia) within the 3 months
* Subject has had any vaccination within 2 weeks prior to Screening or plans to have any vaccination during the study
* Subject has a history of known or suspected intolerance, allergy, or hypersensitivity to olanzapine or opioid antagonists, , or any component of the study drug (eg naltrexone, naloxone)
* Subject has a history of cardiovascular disease, cerebrovascular disease, a seizure disorder, personal or family history of neuroleptic malignant syndrome, or known risk of narrow-angle glaucoma or orthostatic hypotension
* Subject has a current or anticipated need for prescribed opioid medication during the study period
* Subject has a positive urine drug screen for amphetamine, barbiturates, cannabinoids, cocaine, or opioids or positive cotinine test

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to 48 hours post-dose (AUC0 48) | Up to 15 days
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | Up to 15 days
Area under the concentration-time curve from time zero to infinity (AUC∞) | Up to 15 days
\Maximum observed concentration (Cmax) | Up to 15 days
Time to reach Cmax (tmax) | Up to 15 days
Terminal half-life (t½) | Up to 15 days

SECONDARY OUTCOMES:
Total amount of drug excreted in milk (milligrams) | Up to 15 days
Relative drug excreted in milk to dose percentage | Up to 15 days
Estimated infant dose (mg/kg) | Up to 15 days
Estimated relative infant dose to the weight-adjusted maternal dose (%) | Up to 15 days
Incidence of adverse events | Up to 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Yagoda, MD, PhD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Investigator Site, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No